CLINICAL TRIAL: NCT06165601
Title: Evolution of Proteinuria in Renal Transplant Patients Treated with Dapagliflozin for Nephroprotection. DAPAGREFFE
Brief Title: Proteinuria in Renal Transplant Patients Treated with Dapagliflozin
Acronym: DAPAGREFFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL23_0102; 2023-506295-26-00 (Other: EMA)
Record Dates: First submitted 2023-11-20; First posted 2023-12-11 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dapagliflozine (Other): For prospective cohort, an additional follow-up at D14 and M1 will be carried out.
  Interventions: Procedure: Follow-up at D14; Procedure: Follow-up at M1

INTERVENTIONS:
Procedure: Follow-up at D14 — A blood test and urinary test will be performed at D14.
Procedure: Follow-up at M1 — A blood test and urinary test will be performed at M1.

SUMMARY:
The prevalence of chronic kidney disease is rising steadily and represents a major public health challenge. Hypertension and proteinuria are two factors strongly associated with the progression of chronic kidney disease (CKD) and the high risk of cardiovascular complications. Achieving blood pressure control and reducing proteinuria is therefore a major objective in the management of chronic renal failure. Until recently, inhibitors of the renin-angiotensin-aldosterone system were the only therapeutic class known to have both anti-proteinuric and anti-hypertensive action, reducing the risk of progression to end-stage renal disease.

The Investigators intend to conduct an observational study with the primary objective of studying the evolution of proteinuria in kidney transplant patients treated with dapagliflozin according to the marketing authorization. The secondary objectives of the study are to investigate other expected benefits, including effects on renal function and metabolic effects, as well as potential side-effects of this treatment in this population.

DETAILED DESCRIPTION:
Recent years have seen the emergence of sodium-glucose co-transporter type 2 (SGLT2) inhibitors, also known as gliflozins, which represent a real therapeutic innovation in the management of type 2 diabetes, heart failure and chronic kidney disease.

The prevalence of chronic kidney disease is rising steadily and represents a major public health challenge. Hypertension and proteinuria are two factors strongly associated with the progression of chronic kidney disease (CKD) and the high risk of cardiovascular complications. Achieving blood pressure control and reducing proteinuria is therefore a major objective in the management of chronic renal failure. Until recently, inhibitors of the renin-angiotensin-aldosterone system were the only therapeutic class known to have both anti-proteinuric and anti-hypertensive action, reducing the risk of progression to end-stage renal disease.

Several large international studies, initially investigating the efficacy of SGLT2 inhibitors as anti-diabetic therapy, reported that this new therapeutic class reduced the risk of cardiovascular complications and end-stage renal disease. This nephroprotective and cardioprotective effect was independent of the anti-diabetic effect of the drug. The nephroprotective effect is explained in particular by a decrease in proteinuria via a reduction in glomerular hyperfiltration, and a reduction in intraglomerular pressure via vasoconstriction of the afferent artery in response to the blockade of glucose and sodium reabsorption in the proximal convoluted tubule.

An international study (Dapagliflozin and Prevention of Adverse Outcomes in Chronic Kidney Disease study) was specifically designed to investigate the nephroprotective effect of dapagliflozin in both diabetic and non-diabetic proteinuric CKD patients. This study, which included 4,300 patients with glomerular filtration rate (GFR) between 25 and 75ml/min/1.73m2 and an albuminuria/creatinuria ratio between 200 and 5,000mg/g, confirmed a significant reduction in proteinuria, a lower risk of progression to end-stage CKD and a lower mortality rate in patients treated with dapagliflozin compared with those who received placebo. Following this study, Dapagliflozin was granted marketing authorization in France in October 2021 for any patient with chronic kidney disease, in patients with a GFR between 25 and 75ml/min/1.73m2 and an albuminuria/creatinuria ratio between 200 and 5000mg/g despite treatment with converting enzyme inhibitor/Angiotensin II receptor antagonists for at least 4 weeks. Renal transplantation is not a contraindication to the use of dapagliflozin, so renal transplant patients meeting these same criteria may receive dapagliflozin as nephroprotective therapy. However, few data are currently available on the evolution of proteinuria and GFR in this population.

After renal transplantation, proteinuria is also a major factor associated with impaired graft function and cardiovascular risk. However, transplant patients have specific characteristics compared with non-transplant CKD patients: by definition, they have a single functional kidney and receive immunosuppressive treatments that modify renal hemodynamics, including calcineurin inhibitors, drugs that also have a vasoconstrictive effect. In addition, a moderate increase in the risk of urinary tract infection and genital mycotic infection has been reported with the use of gliflozins, necessitating careful monitoring of the incidence of these side effects in this population.

The investigators have been progressively introducing the use of dapagliflozin as a nephroprotective treatment in transplant patients meeting marketing authorisation criteria (chronic renal failure with GFR between 25-75ml/min/1.73m2, albuminuria/creatinuria ratio 200-5000mg/g despite treatment with converting enzyme inhibitors and Angiotensin II receptor antagonists for at least 4 weeks) within the nephrology department of Montpellier University Hospital for several months. To date, more than 30 transplant patients have been treated with dapagliflozin (of whom 12 treated patients have usable data and may be included retrospectively in this study). In this recent experience, a very good safety profile was observed and no drug interactions were identified. Although a reduction in early proteinuria was observed, the follow-up of these patients is not yet long enough to carry out a preliminary analysis.

The investigators intend to conduct an observational study with the primary objective of studying the evolution of proteinuria in kidney transplant patients treated with dapagliflozin according to marketing authorization criteria. The secondary objectives of the study are to investigate other expected benefits, including effects on renal function and metabolic effects, as well as potential side-effects of this treatment in this population.

ELIGIBILITY:
Inclusion Criteria:

* Initiation of dapagliflozin less than 14 days ago for chronic kidney disease
* Glomerular Filtration Rate (GFR) (by CKD-EPI) between 25 and 75 ml.min.1.73m².
* Albuminuria/Creatinuria ratio between 200 mg/g and 5000 mg/g
* Treatment with an ACE inhibitor or angiotensin 2 receptor blocker (ARA II or sartan) at the maximum tolerated dose for at least 4 weeks.
* Age ≥ 18 years

Exclusion Criteria:

* For study group (CKD Renal transplant recipients) : Renal transplantation < 1 year old
* For the control group (non-transplanted CKD) : history of transplantation of an other organ than a kidney initiation or modification of immunosuppressive therapy less than 6 months ago (except temporary discontinuation for infection or change in dosage)
* Type 1 diabetes
* Severe liver failure (Child-Pugh stage C)
* Intolerance to any of the excipients of Forxiga®, in particular lactose intolerance
* Patient undergoing treatment with another SGLT2 inhibitor (sodium-glucose co-transporter type 2)
* Patient enrolled in another clinical trial
* Pregnancy or breast-feeding
* Guardianship or trusteeship
* Patient protected by law
* Subject not affiliated to a social security scheme, or not benefiting from such a scheme
* Patient deprived of liberty
* For the retrospective cohort: Patient's refusal to take part in the study after receiving the information note.
* For the prospective cohort: Failure to obtain written informed consent after a period of reflection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in albuminuria/creatinuria ratio at 6 months | From baseline to 6 months
  decrease in albuminuria/creatinuria ratio ≥ 50% from baseline or achievement of albuminuria/creatinuria ratio ≤ 30 mg/g

SECONDARY OUTCOMES:
Change in albuminuria/creatinuria ratio at 3 months | From baseline to 3 months
  decrease in albuminuria/creatinuria ratio ≥ 50% from baseline or achievement of albuminuria/creatinuria ratio ≤ 30 mg/g
Change in glomerular filtration rate (GFR) | From baseline to 3 and 6 months
  Decrease ≥ 50% in glomerular filtration rate (GFR) from baseline to M3 and M6
Number of patients with end-stage chronic kidney disease (CKD) | From baseline to 3 and 6 months
  Number of patients with end-stage CKD as defined by dialysis or pre-emptive transplant replacement therapy
Number of episodes of acute renal failure | From baseline to 3 and 6 months
  Numbers of episodes of acute renal failure defined according to KDIGO criteria (stage I: increase in serum creatinine ≥ 26.52 micromoles/L in 48 hours or increase in serum creatinine of ≥ 1.5 times the initial value in the preceding 7 days, stage II: increase in serum creatinine ≥ 2 times the initial value, stage III: increase in serum creatinine ≥ 3 times the initial value or serum creatinine ≥ 353. 6 mmol/l or need to start extrarenal purification
Death rate | From baseline to 3 and 6 months
  Death rate from any cause
Study of interaction with immunosuppressive treatments | From baseline to 3 and 6 months
  Study of interaction with immunosuppressive treatments (residual rate and change in dosage of immunosuppressive treatment)
Changes in blood pressure | From baseline to 3 and 6 months
  Systolic blood pressure and diastolic blood pressure are measured in Mmhg
Changes in weight | From baseline to 3 and 6 months
  Weight is measured in kg.
Changes in Hba1c | From baseline to 3 and 6 months
  The dosage of glycated hemoglobin is expressed as a percentage.
Occurrence of infectious side effects | From baseline to 3 and 6 months
  Occurrence of infectious side effects, including urinary tract infections, genital mycotic infections, Fournier's gangrene at M3 and M6
Occurrence of metabolic side effects | From baseline to 3 and 6 months
  Occurrence of metabolic side effects including diabetic ketoacidosis, hypoglycemia, dehydration, hypotension, hydrosodium depletion at M3 and M6
Other adverse reactions associated with dapagliflozin at M3 and M6 | From baseline to 3 and 6 months
  Other adverse reactions : non-infectious and non-metabolic associated with dapagliflozin at M3 and M6
Discontinuation of treatment for side effects | From baseline to 3 and 6 months
  Discontinuation of treatment for side effects

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, France